CLINICAL TRIAL: NCT06933329
Title: Phase 2 Study of Zelenectide Pevedotin in Participants With Previously-Treated NECTIN4 Amplified Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Zelenectide Pevedotin in NECTIN4 Amplified Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BicycleTx Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT8009-202 (Duravelo-4)
Record Dates: First submitted 2025-04-16; First posted 2025-04-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NECTIN4; Zelenectide pevedotin; Advanced or Metastatic; NSCLC; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (non-squamous NSCLC) (Experimental)
  Interventions: Drug: Zelenectide pevedotin (BT8009)
- Cohort B (squamous NSCLC) (Experimental)
  Interventions: Drug: Zelenectide pevedotin (BT8009)

INTERVENTIONS:
Drug: Zelenectide pevedotin (BT8009) — Participants will receive zelenectide pevedotin on Days 1, and 8 of every 21-day cycle.

SUMMARY:
This is a global, multicenter, open-label study that aims to assess the efficacy and safety of zelenectide pevedotin in participants with previously treated NECTIN4-amplified advanced or metastatic non-small cell lung cancer (NSCLC) who have received at least one line of therapy in the advanced/metastatic setting (see inclusion criteria below). The study will comprise of 2 cohorts: Cohort A (non-squamous NSCLC) and Cohort B (squamous NSCLC).

ELIGIBILITY:
Key Inclusion Criteria

* Histologically or cytologically confirmed advanced or metastatic NSCLC.

  1. Cohort A: Histologically or cytologically confirmed non-squamous NSCLC.
  2. Cohort B: Histologically or cytologically confirmed squamous NSCLC.
* Confirmed NECTIN4 gene amplification by an analytically validated clinical trial assay.
* Participants must not have received more than 3 prior lines of systemic therapy in the advanced/metastatic setting.

  * Participants with no known actionable genomic alterations must have received both platinum based therapy and immunotherapy given either sequentially or in combination for advanced/metastatic NSCLC.
  * Those with known actionable genomic alterations (eg, EGFR, ALK, BRAF, MET, ROS1, NTRK1/2/3, RET) are eligible provided they have received or are not candidates for available standard targeted therapy in the advanced/metastatic setting.
* Measurable disease as defined by RECIST v1.1.
* Adequate archival or fresh tumor tissue comprised of advanced or metastatic NSCLC should be available for submission to central laboratory, if not provided during prescreening.
* Life expectancy ≥ 12 weeks.
* Eastern Cooperative Oncology Group Performance Status of ≤ 1.

Key Exclusion Criteria

* Evidence of mixed small cell lung cancer (SCLC) and NSCLC histology.
* Prior treatment with monomethyl auristatin E (MMAE) (vedotin) based therapy.
* Known hypersensitivity or allergy to any of the ingredients of any of the study interventions, or to MMAE.
* Ongoing clinically significant toxicity (Grade ≥ 2) associated with prior treatment for NSCLC (including radiotherapy or surgery), with the exception of well-controlled immuno-oncology related endocrine disorders on supportive or replacement therapy, and alopecia.
* Active keratitis or corneal ulcerations.
* Active or untreated central nervous system (CNS) metastases.
* Uncontrolled diabetes or hypertension.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent draining procedures (monthly or more frequently).
* Active interstitial lung disease or pneumonitis requiring ongoing treatment with steroids (>10mg/day of prednisone or equivalent) or other immunosuppressive medications; or any prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids.
* History or another active malignancy that would interfere with the safety or efficacy evaluation of the clinical study.
* Requirement, while on study, for treatment with strong inhibitors or strong inducers of human cytochrome P450 3A ([cytochrome P450 3A] CYP3A) or inhibitors of P-glycoprotein (P-gp) including herbal- or food-based inhibitors.
* Prior treatment with any systemic anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to first dose of study treatment.

Note: Additional protocol defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) as assessed by Investigator | Up to approximately 3 years
  Percentage of participants with either a confirmed complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Number of participants reporting adverse events (AEs) and abnormalities in laboratory, electrocardiogram (ECG) and vital signs | Up to approximately 3 years
  Safety will be reported as incidence of treatment-emergent adverse events using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 criteria.
Duration of Response (DOR) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  DoR as measured by the time from first documentation of objective response to the first documentation of disease progression or to death (due to any cause), whichever occurs first.
Disease Control Rate (DCR) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  Percentage of participants with confirmed CR, PR, or stable disease (SD)
Clinical Benefit Rate (CBR) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  Percentage of participants with CR, PR or SD ≥16 weeks
Progression Free Survival (PFS) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  PFS is measured by the time from the first day of study drug administration (Day 1) to the first documentation of disease progression, or to death (due to any cause), whichever occurs first.
Overall Survival (OS) | Up to approximately 3 years
  OS is defined as length of time from the first day of study drug administration (Day 1) to death (due to any cause).
Time to Progression (TTP) per RECIST v1.1 as assessed by the Investigator | Up to approximately 3 years
  TTP is defined as the time from first dose of study drug administration until first documentation of disease progression

CONTACTS AND LOCATIONS:
Locations (25):
- United States (10):
  - Alaska Oncology and Hematology, LLC, Anchorage, Alaska
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - St. Vincent Regional Hospital - Cancer Centers of Montana, Billings, Montana
  - Clinical Research Alliance, Inc, Westbury, New York
  - Oncology Hematology Care Clinical Trials, LLC, Fairfield, Ohio
  - Texas Oncology - Central South, Austin, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Virginia Cancer Specialists, Arlington, Virginia
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Leon Berard, Lyon
  - Hopital Foch, Suresnes
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Regional Universitatio (Hospital Civil), Málaga
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clinico Universitatio Lozano Blesa, Zaragoza
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham (University Hospitals Birmingham NHS Foundation Trust), Birmingham
  - University College London Hospital, London
  - The Royal Marsden Hospital, London
  - Northern Centre for Cancer Care, Freeman Hospital (The Newcastle upon Tyne Hospitals NHS Foundation Trust), Newcastle
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No